CLINICAL TRIAL: NCT05164549
Title: Extended-release Pharmacotherapy for Opioid Use Disorder (EXPO): Protocol for an Open-label Randomised Controlled Trial of Injectable Maintenance Buprenorphine With Personalised Psychosocial Intervention.
Brief Title: Extended-release Pharmacotherapy for Opioid Use Disorder
Acronym: EXPO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other); Greater Manchester Mental Health NHS Foundation Trust (Other); Northumberland, Tyne and Wear NHS Foundation Trust (Other); Birmingham and Solihull Mental Health NHS Foundation Trust (Other); NHS Tayside (Other Government); Bangor University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 255522
Record Dates: First submitted 2021-10-27; First posted 2021-12-20 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2021-10

CONDITIONS: Opiate Substitution Treatment
Keywords: opiate; opioid; opioid treatment
MeSH Terms: interventions — Sublocade; Methadone; Buprenorphine; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- XR-Bup (Experimental): Extended-Release Buprenorphine, monthly, 300mg or 100mg
  Interventions: Drug: Buprenorphine Injectable Product
- Bup/Met (Active Comparator): Standard of Care; either Buprenorphine (including Subutex, Suboxone & Espranor) or Methadone (Participant Preference).
  Interventions: Drug: Methadone; Drug: Buprenorphine
- XR-Bup + PSI (Experimental): Extended-Release Buprenorphine, monthly, 300mg or 100mg + Personalised Psychosocial Intervention (PSI)
  Interventions: Drug: Buprenorphine Injectable Product
- Bup/Met + PSI (Active Comparator): Standard of Care; either Buprenorphine (including Subutex, Suboxone & Espranor) or Methadone (Participant Preference) + Personalised Psychosocial Intervention (PSI)
  Interventions: Drug: Methadone; Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine Injectable Product — Investigational Medicinal Product
  Other Names: Sublocade®; prev. RBP-60000
  Arms: XR-Bup; XR-Bup + PSI
Drug: Methadone — Standard of Care
  Arms: Bup/Met; Bup/Met + PSI
Drug: Buprenorphine — Standard of Care
  Other Names: Suboxone; Espranor; Subutex
  Arms: Bup/Met; Bup/Met + PSI

SUMMARY:
The primary objective is a clinical superiority effectiveness contrast to standard of care. Reported following SPIRIT and CONSORT standards, the study will determine whether extended-release injectable depot Buprenorphine (XR-Bup) maintenance therapy for OUD over six months is clinically superior to standard-of-care, oral medication (sublingual Buprenorphine [SL-Bup] or oral methadone [Met]; together: Bup/Met)

DETAILED DESCRIPTION:
EXPO is a pragmatic, multi-centre, open label, four-arm, parallel group, superiority RCT, with a qualitative (mixed-methods) evaluation. The objective of the study is to determine the effectiveness and cost-effectiveness of XR-BUP versus SOC SL-BUP or MET. The primary study endpoint is six months of study treatment. EXPO also contains a single-site evaluation of the effectiveness of XR-BUP with adjunctive PSI versus SOC with adjunctive PSI. Participants allocated to XR-BUP can request to receive longer-term treatment for the duration of the study.

The study population is adults (≥18 years) enrolled in standard-of-care medication treatment for OUD. The study setting is specialist community addiction treatment programmes operated by the National Health Service in England and Scotland. There will be five participant treatment sites in South-East England (South London); North-East England (Newcastle); West Midlands, England (Solihull and Wolverhampton); North-West England (Manchester), and Tayside, Scotland (Dundee).

Groups

In all sites, participants will be randomly allocated to one of two groups:

Group 1. Injectable medication for OUD for 24 weeks (XR-BUP; the experimental condition) Group 2. Oral medication for OUD for 24 weeks (SL-BUP or MET; the control condition).

At the EXPO co-ordinating centre in South London, there will also be random allocation of participants to two additional groups, as follows:

Group 3. Injectable medication for OUD with adjunctive PSI for 24 weeks (XR-BUP with PSI; the experimental condition)

Group 4. Oral medication for OUD with adjunctive PSI for 24 weeks (SL-BUP or MET with PSI; the control condition).

Study aims

Across 24-weeks of study treatment, the primary aim of the EXPO study is to determine:

1. The effectiveness and cost-effectiveness of XR-BUP versus SL-BUP or MET; and
2. The effectiveness of XR-BUP with PSI versus SL-BUP or MET with PSI.

Across 24-weeks of study treatment, secondary study aims will determine the:

1. Safety of XR-BUP;
2. Retention of XR-BUP; SL-BUP; MET; XR-BUP with PSI; and SL-BUP or MET with PSI;
3. Effectiveness of XR-BUP and SL-BUP and MET to reduce opioid craving;
4. Effectiveness of XR-BUP; SL-BUP; MET; XR-BUP with PSI; SL-BUP with PSI; and MET with PSI to reduce use of heroin, cocaine, and benzodiazepines;
5. Effectiveness of XR-BUP and SL-BUP and MET to improve social functioning and recovery.
6. Cost-effectiveness of XR-BUP versus SL-BUP and MET, based on the incremental cost per quality-adjusted life year (QALY) gained.

Study aims will be evaluated by following a pre-registered statistical and health economic analysis plan.

ELIGIBILITY:
IInclusion criteria

1. Aged ≥ 18 years (no upper age limit);
2. Current diagnosis of DSM-5 OUD via SCID-5-RV (moderate-severe at baseline for current episode);
3. Currently enrolled on Met (30mg/day or less) or sublingual Bup or Bup-NX (24mg/day or less) or Esp (18mg/day or less) and in the view of the clinician would be able to convert to XR-Bup within 7 days post randomisation;
4. Voluntarily seeking treatment and able to attend the clinic as required in the protocol;
5. Able to communicate in English to level required to accept standard care and psychosocial intervention;
6. Possession of a contactable personal mobile phone or landline telephone number and ability to nominate at least one locator individual with a verifiable address and a telephone number to assist with the arrangement of follow-up appointments;
7. Living circumstances judged to be of sufficient stability to be able to engage/adhere to the study protocol;
8. Is not pregnant (confirmed) or breast feeding and, if currently or intending to have potentially procreative intercourse, agrees to use a birth control method (either oral hormonal contraceptives, barrier [condom or diaphragm], or Nexplanon implant) for the duration of the study.

8.2 Exclusion criteria

1. Clinically significant medical condition or observed abnormalities on physical examination or laboratory investigation, including but not limited to:

   1. uncontrolled hypertension, significant heart disease (including angina and myocardial infarction in past 12 months), or any cardiovascular abnormality which is judged to be clinically significant;
   2. severe alcohol dependence/withdrawal syndrome which is judged to be clinically significant and may constitute a risk to the patient's safety;
   3. acute hepatitis taken as clinical jaundice on examination, or evidence of blood bilirubin level above the normal range for local reference criteria, or evidence of serum levels of aspartate aminotransferase, alanine aminotransferase levels that are more than three-times the upper limit of the normal range;
2. History of allergic or adverse reactions to Bup or the proprietary ATRIGEL delivery system for XR-Bup (Sublocade®)*;
3. Clinically significant or uncontrolled mental health problems (including but not limited to psychosis, bipolar disorder, schizoaffective disorder), or history or evidence of organic brain disease or dementia that may compromise safety or compliance with the study protocol;
4. Current (past 30 day) suicide plan or suicide attempt in past six months;
5. Current criminal justice involvement with legal proceedings, which in the opinion of a medically qualified investigator indicates a risk that the patient would fail to complete the study protocol due to re-incarceration or move away from the centre's catchment area.
6. Currently taking oral or depot naltrexone therapy or enrolment in any form of naltrexone therapy within 90 days prior to study screening;
7. Any contraindication to Bup*.

   * Participant is ineligible if they have any allergic or adverse reactions or contraindication to Buprenorphine. If participant has any allergic or adverse reaction or contraindication to Met or naloxone, or excipients of Bup-NX or Esp they can be prescribed Bup within the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Count of days abstinent From illicit/non-medical opioids during weeks 2 to 24 (range: 0-161 days) | 24 weeks
  Combining self-report information from Time-Line Follow-Back interview adapted from the Treatment Outcomes Profile and incorporating data from 12 scheduled urine drug screens.

SECONDARY OUTCOMES:
Clinical superiority of XR-Bup plus PSI versus Bup/Met plus PSI | 24 weeks
  Number of days abstinent from cocaine Days 8 - 168 Number of days abstinent from Benzodiazepines Days 8 - 168 Longest time in days continuously abstinent from heroin Days 8 - 168 Longest time in days continuously abstinent from cocaine Days 8 - 168 Longest time in days continuously abstinent from Benzodiazepines Days 8 - 168
Cost-effectiveness of XR-BUP versus Bup and Met | 24 weeks
  Based on the incremental cost per quality-adjusted life year (QALY) gained.
Safety of XR-Bup | 24 weeks
  Number of safety events from study enrolment to 24 weeks
Time (days) enrolled in study treatment (retention) to week 24 | 24 weeks
OUD remission status (DSM5 OUD severity; SCID-5-RV) | 24 weeks
Clinician rating of severity, complexity and recovery strengths: ADAPT | 24 weeks
Clinician global impression of severity and improvement): CGI-S/I; | 24 weeks
Count of days abstinent from cocaine and illicit/non-medical benzodiazepines | 24 weeks
  During weeks 2 to 24 (range: 0-161 days); combining self-report information from Time-Line Follow-Back interview adapted from the Treatment Outcomes Profile and incorporating data from 12 scheduled urine drug screens
Frequency of opioid (H) and cocaine (C) craving experience: CEQ-F(H) and CEQ-F(C) | 24 weeks
Craving need and want strength for heroin and cocaine: VAS-N(H/C) and VAS-W(H/C) | 24 weeks
Difficulties in Emotion Regulation (Short Form): DERS-SF | 24 weeks
Depression symptoms: QIDS-SR | 24 weeks
Work and social adjustment: WSAS | 24 weeks
Subjective recovery and improvement: SURE | 24 weeks
Patient rating of OUD severity and improvement: | 24 weeks
  Utilising PRO-S/I;
Patient rating of OUD severity and improvement: | 24 weeks
  Cognitive impairment: MoCA
Alcohol consumption: typical quantity and frequency: (ALC-QFM) | 24 weeks
Longer Term Outcomes | Through study completion, up to 4 years
  Among participants enrolled in longer term XR-BUP treatment: heroin, cocaine and illicit/non-medical benzodiazepine use in past 90 days (TLFB; UDS)
Longer Term Outcomes | Through study completion, up to 4 years
  Among participants enrolled in longer term XR-BUP treatment: OUD and CUD remission status (SCID-5-RV)
Longer Term Outcomes | Through study completion, up to 4 years
  Among participants enrolled in longer term XR-BUP treatment: somatic symptoms (PHQ-15)
Longer Term Outcomes | Through study completion, up to 4 years
  Among participants enrolled in longer term XR-BUP treatment: emotion regulation (DERS-SF)
Longer Term Outcomes | Through study completion, up to 4 years
  Among participants enrolled in longer term XR-BUP treatment: depression and anxiety symptoms (PHQ-4)
Longer Term Outcomes | Through study completion, up to 4 years
  Among participants enrolled in longer term XR-BUP treatment: quality of life (OSTQOL)

CONTACTS AND LOCATIONS:
Overall Officials: Mike Kelleher, Dr, Principal Investigator — South London and Maudsley NHS Foundation Trust
Locations (5):
- United Kingdom (5):
  - Birmingham and Solihull Mental Health NHS Foundation Trust, Birmingham
  - NHS Tayside, Dundee
  - South London and Maudsley NHS Foundation Trust, London
  - Greater Manchester Mental Health NHS Foundation Trust, Manchester
  - Cumbria, Northumberland, Tyne and Wear NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marsden J, Kelleher M, Hoare Z, Hughes D, Bisla J, Cape A, Cowden F, Day E, Dewhurst J, Evans R, Hearn A, Kelly J, Lowry N, McCusker M, Murphy C, Murray R, Myton T, Quarshie S, Scott G, Turner S, Vanderwaal R, Wareham A, Gilvarry E, Mitcheson L. Extended-release pharmacotherapy for opioid use disorder (EXPO): protocol for an open-label randomised controlled trial of the effectiveness and cost-effectiveness of injectable buprenorphine versus sublingual tablet buprenorphine and oral liquid methadone. Trials. 2022 Aug 19;23(1):697. doi: 10.1186/s13063-022-06595-0. PMID 35986418
- [Result] Marsden J, Kelleher M, Gilvarry E, Mitcheson L, Bisla J, Cape A, Cowden F, Day E, Dewhurst J, Evans R, Hardy W, Hearn A, Kelly J, Lowry N, McCusker M, Murphy C, Murray R, Myton T, Quarshie S, Vanderwaal R, Wareham A, Hughes D, Hoare Z. Superiority and cost-effectiveness of monthly extended-release buprenorphine versus daily standard of care medication: a pragmatic, parallel-group, open-label, multicentre, randomised, controlled, phase 3 trial. EClinicalMedicine. 2023 Nov 17;66:102311. doi: 10.1016/j.eclinm.2023.102311. eCollection 2023 Dec. PMID 38045803
- See also: EXPO Trial Primary Results Publication — https://pubmed.ncbi.nlm.nih.gov/38045803/
- See also: EXPO Trial Protocol — https://pubmed.ncbi.nlm.nih.gov/35986418/

DOCUMENTS (2):
  • Study Protocol (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/49/NCT05164549/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/49/NCT05164549/SAP_001.pdf